CLINICAL TRIAL: NCT07007000
Title: Cardio-neural Pacing to Modulate AV Conduction in Persistent AF Patients - a Feasibility Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tam Tsz Kin, Prof, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNP study
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Cardio-neural Pacing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardio-neural pacing (Other): Patient will undergo temporary cardio-neural pacing during implantation of pacemaker
  Interventions: Device: Temporary cardio-neural pacing

INTERVENTIONS:
Device: Temporary cardio-neural pacing — After routine ventricular lead implantation, a coronary sinus sheath will be delivered to RA septum, posterior to CS ostium, at the expected location of parasympathetic ganglion plexus. Pace mapping will be performed with a pacing lead at 30Hz, variable amplitude (20, 10, 5V) at 1ms pulse width. An electrophysiology catheter may be used where necessary for pace-mapping the response. At the site where lowest output can generate 30% prolongation of ventricular CL, the lead is fixed for 2-5mm depth. The output is tested again to achieve 50% prolongation of ventricular CL (at 20, 10, 5, 2, 1V). Fluoroscopic image will be collected with contrast injection at the sheath. Repositioning of lead can be performed if the rate suppression cannot be achieved with 3V@0.4ms. Implanted lead will serve as an atrial sensing and pacing lead and will not be removed at the end of procedure. Patient will be connected to a dual to a dual chamber pacemaker with device programming per usual clinical care.

SUMMARY:
Atrial fibrillation is the commonest arrhythmia with a lifetime risk of one in 3-5. In patients with late stage of persistent atrial fibrillation, rate control is usually preferred over rhythm control. Besides medication therapy, atrioventricular nodal ablation is sometimes required with placement of a pacemaker afterwards.

The AV node is being innervated by parasympathetic fibres that modulate its conduction. Ablation in these parasympathetic innervations around the coronary sinus (at the CS ostium or posterior to it) has been shown to be promising for treating vagal mediated syncope. Stimulation of these fibres with high frequency pacing could achieve chronic heart rate suppression in animal model. Intermittent pacing in this area has also been shown to be successful in reducing ventricular rate in atrial fibrillation to prevent inappropriate ICD shock.

As a proof-of-concept case, we attempted pacing cardio-neural fibres in one of our patients. Pacing 30Hz at 10mA, 2ms pacing in ostial or postero-septal coronary sinus both resulted in a dose dependent prolongation of VV cycle length during atrial fibrillation. Patient did not complain of discomfort during such pacing. We postulate that pacing these fibers can achieve rate control and avoid the need for rate control medication or AV node ablation in some of these patients.

This study aims to evaluate safety and efficacy of temporary cardio-neural pacing (CNP), and collect fluoroscopic images and electroanatomical mapping data on cardio-neural pacing sites.

DETAILED DESCRIPTION:
This is a prospective cohort study. 10 patients with persistent atrial fibrillation with pacing indication will be recruited. They are all scheduled to undergo permanent transvenous pacemakers according to clinical need. Informed consent will be signed before procedure. Arterial line will be inserted for monitoring of blood pressure. After routine ventricular lead implantation, a coronary sinus sheath (attain command or deflectable) will be delivered to RA septum, posterior to CS ostium, at the expected location of parasympathetic ganglion plexus. Pace mapping will be performed with a pacing lead (such as Select Secure 3830) at 30Hz, variable amplitude (20, 10, 5V) at 1ms pulse width. An electrophysiology catheter may be used where necessary for pace-mapping the response. At the site where lowest output can generate 30% prolongation of ventricular CL, the lead is fixed for 2-5mm depth. The output is tested again to achieve 50% prolongation of ventricular CL (at 20, 10, 5, 2, 1V). Fluoroscopic image will be collected with contrast injection at the sheath. Repositioning of lead can be performed if the rate suppression cannot be achieved with 3V@0.4ms. Eventually, the implanted lead will serve as an atrial sensing and pacing lead and will not be removed at the end of procedure. Patient will be connected to a dual chamber pacemaker with device programming per usual clinical care. Patients will be followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent atrial fibrillation who are scheduled for pacemaker implantation per guideline indication

Exclusion Criteria:

* Patients who cannot provide informed consent
* Patients < 18 years old
* Pregnant patients
* Illiterate patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percentage prolongation of CL | In implant procedure
  Measure percentage prolongation of CL with lead fixation

SECONDARY OUTCOMES:
Threshold | In implant procedure
  Determine the lowest threshold to achieve prolongation
Discomfort | In implant procedure
  Any discomfort from patient during cardio-neural pacing
Average arterial line blood pressure | In implant procedure
  Evaluate average arterial line blood pressure during cardio-neural pacing, compared with that before the pacing.
Fluoroscopic imaging | In implant procedure
  Collect fluoroscopic imaging to identify location and range of anatomical target area

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong